CLINICAL TRIAL: NCT02582450
Title: Validation of a Specific Measure for Assessment of Compliance With Treatment in Patients With Hemophilia. Veritas-Pro Project
Brief Title: Validation of a Specific Measure for Assessment of Compliance With Treatment in Patients With Hemophilia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Real Fundación Victoria Eugenia (Other)
Collaborators: Medtep Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Veritas-Validation
Record Dates: First submitted 2015-10-19; First posted 2015-10-21 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Haemophilia
Keywords: Haemophilia; Adherence of Treatment; Knowledge of Illness; Medical-patient Relationship; Illness Behavior; Treatment Difficulties; Veritas
MeSH Terms: conditions — Hemophilia A; Illness Behavior | interventions — hydroxyethyl methacrylate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with haemophilia: Sample of patients with haemophilia over 18 years of age that will participate in piloting of reliability and validity of the Spanish version of the Veritas-Pro questionnaire.
  Interventions: Other: Patients with haemophilia

INTERVENTIONS:
Other: Patients with haemophilia — Piloting of reliability and validity of the Spanish version of the Veritas-Pro questionnaire.

SUMMARY:
Research project for validation of a questionnaire on compliance to treatment in patients with hemophilia. It is intended to validate the American VERITAS-PRO scale according to the international methodology validation questionnaires: reverse translation, according to intersubject patients, psychometric validation and reliability analysis with large sample of patients.

DETAILED DESCRIPTION:
The validated questionnaire obtained in this project will identify the actual degree of patient compliance to drug therapy, using as gold standard the difference between the treatment prescribed and administered.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hemophilia A and B
* Patients who have previously signed the informed consent document

Exclusion Criteria:

* Patients with other congenital coaghulopatías (eg, Von Willebrand's disease)
* Patients with cognitive impairment, or oral or written understanding

Ages: 13 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with haemophilia around the country that will participate in study.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2015-09; Primary Completion 2015-10 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Translation of the original questionnaire (English) to Spanish | 1 day (Screening visit)
  Three health experienced in the treatment of hemophilia and knowledge of English, translated into Spanish the HAL and HEP questionnaire. Two native speakers (English and Spanish), reverse-translate the original text of the HAL and HEP questionnaires and the text translated by the Spanish health.
The translated version of the questionnaire | 1 day (Screening visit)
  10 patients with hemophilia adults enrolled randomly will participate in the pilotage.
  The clarity of the questions in Spanish translated version and the relevance of each of the items of the questionnaires will be evaluated.
Sending the questionnaire to a large sample of patients for final validation | 1 day (Screening visit)
  70 patients with hemophilia will participate in the pilotage. The validity and reliability of the Spanish version translated from the questionnaires will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, PhD, Principal Investigator — Real Fundación Victoria Eugenia
Locations (1):
- Real Fundación Victoria Eugenia, Madrid, Madrid, Spain